CLINICAL TRIAL: NCT06454981
Title: Clinical Trial for Effectiveness and Safety Evaluation of Hemodiafilter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Kaiyuan Suixi Medical Technology Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH202101
Record Dates: First submitted 2024-05-17; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Renal Failure Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXCLEAR 800 (Experimental): "Hemodiafilter" (Model & spec.: EXCLEAR 800) produced by Shinva Medical Instrument Co.,Ltd.
  Interventions: Device: Hemodiafilter
- FX 800HDF (Active Comparator): Hollow fibre hemodialysis/filter FX 800HDF (registration certificate no.: GuoMeZhiJin 20193101929) manufactured by Fresenius Medical Care AG & Co.KGaA (Registered agent: Fresenius Medical Care (shanghai) Company Limted)
  Interventions: Device: Fresenius Medical Care AG & Co.KGaA

INTERVENTIONS:
Device: Hemodiafilter — The enrolled patients were randomly divided into the experimental group and the control group, using the "hemodiafilter" (experimental device) produced by Shinva Medical Instrument Co.,Ltd.
  Other Names: EXCLEAR 800
  Arms: EXCLEAR 800
Device: Fresenius Medical Care AG & Co.KGaA — The enrolled patients were randomly divided into the experimental group and the control group, using the FX 800HDF hollow fiber hemodialysis/filter (control device) produced by Fresenius Medical Care AG & Co.KGaA (registered agent: Fresenius Medical Care (shanghai) Company Limted).
  Other Names: FX 800HDF
  Arms: FX 800HDF

SUMMARY:
The clinical trial was conducted in the nephrology department of Shulan (Hang Zhou) Hospital,the hemodialysis room of Wenzhou TCM Hospital, Jinhua Municipal Centeral Hospital, and Tongde Hospital of Zhejiang Province. The clinical trial is designed as a multi-center, randomized, open, positive parallel control, non-inferiority clinical trial. The control devices were positive devices approved by CFDA, which have been widely used and have been proven efficacy for the corresponding indications. The objective of the non-inferiority test is to show that the therapeutic effect of the experimental device is clinically non-inferior to that of the positive control device.

The enrolled patients were randomly divided into the experimental group and the control group, using the "hemodiafilter" (experimental device) produced by Shinva Medical Instrument Co.,Ltd. and the FX 800HDF hollow fiber hemodialysis/filter (control device) produced by Fresenius Medical Care AG & Co.KGaA (registered agent: Fresenius Medical Care (shanghai) Company Limted), respectively. To evaluate the effectiveness, safety and operability of the "hemodiafilter" produced by Shinva Medical Instrument Co.,Ltd. by means of control.Cases were screened according to the inclusion and exclusion criteria. The selected cases were randomised into groups in chronological order.

Based on the principle of voluntary participation of subjects in clinical trial, before the commencement of the clinical trial, the purpose, process and duration of the clinical trial were explained in detail to the subjects, as well as the role of the subjects in using the experimental device on the clinic and the possible risks encountered and the measures to be taken, and the clinical trial was carried out after obtaining the consent of the subjects and signing the Informed Consent Form. The Informed Consent Form was not listed in the report in order to protect the subject's privacy because it was signed by the subject. And it was kept as original information in the clinical trial unit.

The clinical trial protocol and informed consent form had been approved by the ethics committee prior to the clinical trial.

DETAILED DESCRIPTION:
Applicant for Medical Device Registration: Shinva Medical Instrument Co., Ltd. Investigators: Zhangfei Shou, Chief Physician (01 Center Shulan (Hang Zhou) Hospital)Weixia Huang, Chief Physician (02 Center Wenzhou TCM Hospital) Jian Huang, Chief Physician (03 Center Jinhua Municipal Centeral Hospital) Liansheng Liu, Chief Physician (04 Center Tongde Hospital of Zhejiang Province) Objective: Main objective: the main objective of this clinical trial is to ensure the safety of the subjects and the scientific validity of the clinical trial in order to evaluate the effectiveness of the experimental medical device hemodiafilter (EXCLEAR 800) in patients with chronic renal failure with stable condition, compared to the control device, hollow fibre hemodialysis/filter (FX 800HDF) produced by Fresenius Medical Care AG & Co.KGaA, and meet the requirements of China medical device regulations.

Secondary objective: to evaluate the safety of the experimental medical device hemodiafilter (EXCLEAR 800) compared to the control device hollow fibre hemodialysis/filter (FX 800HDF) manufactured by Fresenius Medical Care AG & Co.KGaA for hemodiafiltration treatment in patients with stable chronic renal failure.

Trial Design:The clinical trial was conducted in the nephrology department of Shulan (Hang Zhou) Hospital, the hemodialysis room of Wenzhou TCM Hospital, Jinhua Municipal Centeral Hospital, and Tongde Hospital of Zhejiang Province. The clinical trial is a multi-center, randomized, open, positive parallel control, non-inferiority design.Statistical Methods:General principle

1. Statistical description The quantitative indicators will be described by calculating the mean, standard deviation, median, minimum, maximum, lower quartile (Q1), upper quartile (Q3), and the categorical indicators will be described by the number of instances and percentages of each category.
2. Statistical Inference For comparisons of the general conditions of the two groups, the t-test or Wilcoxon rank-sum test was used to compare the quantitative indicators between groups according to the distribution of data. The chi-square test or exact probability method (if the chi-square test was not applicable) was used for categorical indicators, and the Wilcoxon rank-sum test or the CMH test was used for hierarchical data. SAS 9.4 or higher version software was used as the statistical analysis tool for this study, and the corresponding statistical analysis methods were selected after discussion with clinical workers and based on the clinical characteristics of different indicators. All statistical tests were two-sided unless otherwise stated, and a p-value of less than 0.05 (two-sided) was considered statistically significant. Detailed and additional exploratory analyses may be required in addition to the statistical methods listed below, and will be identified in the Study Report and Analysis Plan (SAP).In PPS, the mean creatinine clearance rate of the main indicator was 182.87 in the experimental group and 175.96 in the control group, with a 95% confidence interval [-4.532, 18.348] for the difference between the two groups. The lower bound of the confidence interval was greater than the non inferiority threshold; The main indicator of urea nitrogen clearance rate is 226.60 in the experimental group and 218.92 in the control group. The 95% confidence interval for the difference between the two groups is [-6.268,21.624], and the lower bound of the confidence interval is greater than the non inferiority threshold; The mean decrease rate of main indicators β2-mg micro globulin in the experimental group was 64.87%, while the mean in the control group was 66.06%. The 95% confidence interval for the difference between the two groups was [-5.309,2.930], and the lower bound of the confidence interval was greater than the non inferiority threshold. The main indicators of the experimental group were not inferior to those of the control group.

Groups: Experimental group: "Hemodiafilter" (Model & spec.: EXCLEAR 800) produced by Shinva Medical Instrument Co.,Ltd.

Control group: Hollow fibre hemodialysis/filter FX 800HDF (registration certificate no.: GuoMeZhiJin 20193101929) manufactured by Fresenius Medical Care AG & Co.KGaA (Registered agent: Fresenius Medical Care (shanghai) Company Limted)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years, male or female;
2. Maintenance dialysis patients with stable chronic renal failure who require hemodiafiltration with a hemodiafilter;
3. To maintain a blood flow of 200 ml/min and above during dialysis;
4. Patients agreed to participate in this trial and signed an informed consent form.

Exclusion Criteria:

1. Patients who are mental disorder or unstable condition;
2. The frequency of dialysis treatment is not satisfied: 2-3 times per week for not less than 4 hours each time, maintained for at least three months;
3. Pregnant women, women preparing for pregnancy and lactating;
4. Patients with severe anaemia, infection, malignancy, active bleeding;
5. Patients with severe cardiac, hepatic and pulmonary diseases;
6. Patients with contraindications to dialysis or allergy to any of the components of the hemodiafilter used in this trial;
7. Patients who are underweight (dry weight less than 40kg);
8. Patients who participated in other clinical trials within 30 days before enrollment that could affect the evaluation of this study;
9. Patients who, in the opinion of the investigator, should not be enrolled in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
The creatinine clearance rate of hemodiafilter | Stable dialysis for 60 minutes±1min
  Stable dialysis for 60 minutes, with fixed blood flow and dialysate flow under working conditions, set ultrafiltration rate to 10ml/min, and simultaneously draw blood from the dynamic and static pulse ends of the dialyzer to measure creatinine and calculate clearance rate.
The urea nitrogen clearance rate of hemodiafilter | Stable dialysis for 60 minutes±1min
  Stable dialysis for 60 minutes, with fixed blood flow and dialysate flow under working conditions, set ultrafiltration rate to 10ml/min, and simultaneously draw blood from the dynamic and static pulse ends of the dialyzer to measure creatinine and calculate clearance rate.
β2-MG reduction rate | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  When measuring the decline rate, blood is drawn at the beginning and end of hemodialysis filtration, ultrafiltration is stopped, and blood flow is first reduced to 100ml/min. After stopping the pump, blood is immediately drawn from the subject's body.

SECONDARY OUTCOMES:
Overall blood dialysis filtration creatinine clearance rate | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Ccr=(140﹣age)×weight(kg)/72×Scr(mg/dl)Ccr=(140﹣age)×weight(kg)/72×Scr(mg/dl) Or Ccr=[(140﹣age)×weight(kg)]/[0.818×Scr(umol/L)] Note：Women according to calculation results×0.85
Overall blood dialysis filtration creatinine decrease rate | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Overall blood dialysis filtration creatinine decrease rate（%）=1-(Creatinine after hemodialysis filtration/creatinine before hemodialysis filtration)×100%
Overall blood dialysis filtration urea nitrogen clearance rate（Kt/V） | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Kt/V=-ln(R-0.008×t)+(4-3.5×R ) ×UF/W Formula： Ln：Natural logarithm ； t ：Hemodialysis filtration treatment time (h)； R ：The ratio of BUN after hemodialysis filtration to BUN before hemodialysis filtration； UF：Ultrafiltration capacity (L)； W ：Patient's weight after blood dialysis filtration (kg).
Urea reduction rate（URR） | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Urea reduction rate（URR，%）＝1-(Blood urea concentration after hemodialysis filtration/blood urea concentration before hemodialysis filtration)×100%
Ultrafiltration rate | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Ultrafiltration rate (ml/h)=total water removal amount (ml)/treatment time (h)
Conduct a blood phosphorus test on the blood of subjects before and after hemodialysis filtration to check if the indicators are qualified. | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Qualified: The researcher determined it to be "normal" or "abnormal with no clinical significance".
  Unqualified: The researcher determined that the abnormality has clinical significance.
Perform C-reactive protein testing on the blood of subjects before and after hemodialysis filtration to check if the indicators are qualified. | blood is drawn at the beginning within 30 minutes and end of hemodialysis filtration within 30 minutes
  Qualified: The researcher determined it to be "normal" or "abnormal with no clinical significance".
  Unqualified: The researcher determined that the abnormality has clinical significance.
Conduct blood gas (PO2) tests on the blood of subjects before and 15 minutes after the start of hemodialysis filtration to check if the indicators are qualified. | blood is drawn at the beginning within 30 minutes, 15min±1min and end of hemodialysis filtration within 30 minutes
  Qualified: The researcher determined it to be "normal" or "abnormal with no clinical significance".
  Unqualified: The researcher determined that the abnormality has clinical significance.
Conduct blood gas (PCO2) tests on the blood of subjects before and 15 minutes after the start of hemodialysis filtration to check if the indicators are qualified. | blood is drawn at the beginning within 30 minutes, 15min±1min and end of hemodialysis filtration within 30 minutes
  Qualified: The researcher determined it to be "normal" or "abnormal with no clinical significance".
  Unqualified: The researcher determined that the abnormality has clinical significance.
Conduct blood gas (HCO3-) tests on the blood of subjects before and 15 minutes after the start of hemodialysis filtration to check if the indicators are qualified. | blood is drawn at the beginning within 30 minutes, 15min±1min and end of hemodialysis filtration within 30 minutes
  Qualified: The researcher determined it to be "normal" or "abnormal with no clinical significance".
  Unqualified: The researcher determined that the abnormality has clinical significance.
Conduct blood gas (pH) tests on the blood of subjects before and 15 minutes after the start of hemodialysis filtration to check if the indicators are qualified. | blood is drawn at the beginning within 30 minutes, 15min±1min and end of hemodialysis filtration within 30 minutes
  Qualified: The researcher determined it to be "normal" or "abnormal with no clinical significance".
  Unqualified: The researcher determined that the abnormality has clinical significance.
Rupture of membrane | during Hemodialysis filtration period within 4 hours
  Whether the hemodiafilter breaks the membrane during treatment. Qualified: No membrane rupture occurred in the hemodiafilter during treatment. Unqualified: Membrane rupture of the hemodiafilter occurred during treatment. If the membrane breaks during treatment, the cause and disposal method shall be recorded.
transmembrane pressure | during Hemodialysis filtration period within 4 hours
  During treatment, whether there is a continuous high transmembrane pressure machine alarm, or even can not be used. Qualified: No machine alarm of continuous high transmembrane pressure occurred during treatment.
  Unqualified: During treatment, a continuous high transmembrane pressure machine alarm occurred, which could not even be used. If the transmembrane pressure of the hemodiafiltration is persistently high during treatment, the machine will alarm or even fail to use. The reason and disposal method should be recorded.
anticoagulant performance | during Hemodialysis filtration period within 4 hours
  Hemodiafiltration coagulation degree classification:
  Grade 0: No coagulation or coagulation with several fibers. Grade I: Partial or fascicular coagulation. Grade II: Severe coagulation or coagulation of more than half of fibers. Grade III: During hemodiafiltration, the hemodiafiltration device (transmembrane pressure and/or venous pressure) is significantly increased or the hemodiafiltration device needs to be replaced due to membrane rupture and other reasons. Qualified: The coagulation degree of hemodiafiltration was graded as "Grade 0-Grade I".
  Unqualified: The degree of hemodiafiltration coagulation was graded as "Grade II or above".

CONTACTS AND LOCATIONS:
Overall Officials: Zhangfei Shou, Principal Investigator — Zhejiang Provincial Tongde Hospital
Locations (1):
- Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang, China